CLINICAL TRIAL: NCT03704389
Title: Behavioral Economics Applications to Geriatrics Leveraging EHRs
Acronym: BEAGLE R21
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: University of California, Los Angeles (Other); University of Southern California (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: STU00205722; R21AG057383 (NIH)
Record Dates: First submitted 2018-10-09; First posted 2018-10-12 (Actual); Results first posted 2025-10-07 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-09

CONDITIONS: Prostate Specific Antigen; Asymptomatic Bacteriuria; Type 2 Diabetes Mellitus
Keywords: Geriatrics; Clinical decision support; Behavioral Economics
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Clinical decision support intervention (Experimental): Participating clinicians will receive any of three clinical decision support nudges within the electronic health record when all eligibility criteria are met within a patient's chart.
  Interventions: Behavioral: Clinical decision support

INTERVENTIONS:
Behavioral: Clinical decision support — Clinical decision support nudges within the electronic health record

SUMMARY:
The risks and benefits of many diagnostic approaches and treatments differ for older adults compared to middle aged adults. When diagnostic and therapeutic strategies are misapplied to older adults this can lead to increased morbidity and mortality. Well established examples where clinicians do not often follow best practices in the care of older adults include those identified by the American Geriatrics Society for the Choosing Wisely initiative: 1) testing and treatment for asymptomatic bacteriuria, 2) prostate specific antigen testing in older men without prostate cancer, and 3) overuse of insulin or oral hypoglycemics for type 2 diabetes.

Clinical decision support nudges, informed by social psychology and delivered via electronic health records (EHRs), are promising strategies to reduce the misuse of services in cases where optimal utilization may not be zero but should be well below current practice. These interventions seek to influence conscious and unconscious drivers of clinical decision making, are low cost to implement and disseminate, and can be incorporated into existing delivery systems. In the R21 phase of this Behavioral Economics Applications to Geriatrics Leveraging EHRs (BEAGLE) study, we will: select EHR delivered nudges to address 3 topics of potential misuse in older adults based on the main psychological drivers of overuse identified in interviews with high-using clinicians; develop and pilot test decision support tools within a health systems' EHR to understand technical feasibility, work flow fit, preliminary impact on clinical outcomes, and clinician acceptability; and develop and validate electronic clinical quality measures of potential overuse/misuse related to the care of older adults.

DETAILED DESCRIPTION:
The risks and benefits of many diagnostic approaches and treatments differ for older adults compared to middle aged adults. When diagnostic and therapeutic strategies are misapplied to older adults this can lead to increased morbidity and mortality. Well-established examples where clinicians do not often follow best practices in the care of older adults include those identified by the American Geriatrics Society for the Choosing Wisely initiative: 1) testing and treatment for asymptomatic bacteriuria, 2) prostate specific antigen testing in older men without prostate cancer, and 3) overuse of insulin or oral hypoglycemics for type 2 diabetes. There are several hypotheses as to why clinicians fail to incorporate best evidence into geriatric clinical care. First, they may underestimate downstream harms of testing which seems easy to do (e.g., a urinalysis for a non-specific symptom) or treatment that may be appropriate for younger patients (e.g. intensifying insulin to achieve tight control). Second, clinicians may overweigh the risks of not performing the action (e.g., missing cancer diagnosis, failing to diagnose urinary tract infection (UTI) in a patient presenting without urinary tract symptoms). Third, clinicians may respond to real or perceived social norms (from patients and their families, other clinicians or both) that set expectations to behave in specific ways. Fourth, force of habit may lead clinicians to act in a way similar to how they have done in the past even if current evidence doesn't support it. And fifth, clinicians may overuse a test or treatment to avoid feeling they are expressing an ageist bias toward their patients. Clinical decision support nudges, informed by social psychology and delivered via electronic health records (EHRs), are promising strategies to reduce the misuse of services in cases where optimal utilization may not be zero but should be well below current practice. These interventions seek to influence conscious and unconscious drivers of clinical decision making, are low cost to implement and disseminate, and can be incorporated into existing delivery systems. In the R21 phase of this Behavioral Economics Applications to Geriatrics Leveraging EHRs (BEAGLE) study, we will: select EHR delivered nudges to address 3 topics of potential misuse in older adults based on the main psychological drivers of overuse identified in interviews with high-using clinicians; develop and pilot test decision support tools within a health systems' EHR to understand technical feasibility, work flow fit, preliminary impact on clinical outcomes, and clinician acceptability; and develop and validate electronic clinical quality measures of potential overuse/misuse related to the care of older adults.

ELIGIBILITY:
Inclusion Criteria:

* Northwestern Medicine primary care clinician caring for adults
* Provides informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 664 (Actual)
Dates: Start 2019-01-17 (Actual); Primary Completion 2019-07-17 (Actual); Study Completion 2019-08-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Northwestern Medicine, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All study outcome data are from patients. We report on the n=664 patients who were attributed to a study clinician with a visit during the intervention period that met denominator criteria for an outcome.
Pre-assignment Details: This is a small non-randomized pilot study. This trial enrolled patients with a waiver of informed consent. Clinicians were not enrolled. All outcome data were collected via the electronic health record. This explains why the number of participants started is the same as the number of participants completed.
Groups:
- Clinical Decision Support Intervention: Primary care clinicians will receive any of three clinical decision support nudges within the electronic health record when all eligibility criteria are met within a patient's chart.
  Clinical decision support: Clinical decision support nudges within the electronic health record
Period: Overall Study
Arm/Group | Clinical Decision Support Intervention
Started | 664
Completed | 664 (We collected study data from automated queries of electronic health record data.)
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: We report age and sex for PSA and UA/UC outcome measures. We have not collected sex for patients eligible for diabetes outcome measure.
Groups:
- Clinical Decision Support Intervention: Participating clinicians will receive any of three clinical decision support nudges within the electronic health record when all eligibility criteria are met within a patient's chart.
  Clinical decision support: Clinical decision support nudges within the electronic health record
  Baseline characteristics were not collected from enrolled clinicians.
Arm/Group | Clinical Decision Support Intervention
Number analyzed (Participants) | 664
Age, Categorical [Count of Participants; unit: Participants] — We report baseline characteristics of patients who met denominator criteria for three study outcome measures for pilot clinicians during the six month intervention period.
  Baseline characteristics were not collected from enrolled clinicians.
  Participants
    <=18 years | 0
    Between 18 and 65 years | 0
    >=65 years | 664
Sex: Female, Male [Count of Participants; unit: Participants] — Population: We do not have sex data for patients eligible for the diabetes measure so that is why the number analyzed in this section is smaller than number of participants overall.
  Participants
    number analyzed (Participants) | 538
    Female | 230
    Male | 308
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 664

OUTCOME MEASURES:

1. Primary Outcome: Misuse of Urinalysis or Urine Culture in Older Women
Description: Percentage of women patients aged 65 years and older who underwent a urinalysis and/or urine culture for suspected urinary tract infection (UTI) who did not have genitourinary specific symptoms
Time Frame: 6 months intervention period
Population: Proportion of female patients aged 65 years and older with a primary care encounter who had a urinalysis or urine culture done for non-specific reasons among those with a test done
Measure: Count of Participants; unit: Participants
Groups:
- Clinical Decision Support Intervention: Clinicians will receive any of three clinical decision support nudges within the electronic health record when all eligibility criteria are met within a patient's chart.
  Clinical decision support: Clinical decision support nudges within the electronic health record
Arm/Group | Clinical Decision Support Intervention
Number analyzed (Participants) | 230
Participants | 25

2. Primary Outcome: Prostate-Specific Antigen (PSA) Testing in the Elderly
Description: Percent of male patients seen by participating clinicians 76 and older with no history of prostate cancer who had a PSA test done during the measurement period
Time Frame: 6 month intervention period
Population: Percent of male patients seen by participating clinicians 76 and older with no history of prostate cancer who had a PSA test done during the measurement period
Measure: Count of Participants; unit: Participants
Arm/Group | Clinical Decision Support Intervention
Number analyzed (Participants) | 308
Participants | 13

3. Primary Outcome: Diabetes Overtreatment in the Elderly
Description: Percent of diabetes patients 75 and older treated with insulin or oral hypoglycemic with hemoglobin A1c less than 7.0.
Time Frame: 6 month intervention period
Population: Percent of diabetes patients 75 and older treated with insulin or oral hypoglycemic with hemoglobin A1c less than 7.0.
Measure: Count of Participants; unit: Participants
Arm/Group | Clinical Decision Support Intervention
Number analyzed (Participants) | 126
Participants | 50

ADVERSE EVENTS:
Time Frame: 6 month intervention period
Description: 1) female patients with an emergency department visit or hospitalization with diagnosis of UTI or sepsis following visit with Clinical Decision Support (CDS) exposure and 2) diabetes patients with an emergency department visit or hospitalization for hyperglycemia following a primary care visit with CDS exposure. Number of patients at risk is not equal to all enrolled subjects. Only subgroups of patients receiving CDS are in the denominator for adverse event reporting.
Groups:
- Clinical Decision Support Intervention: This was a small one arm pilot study. The study had clinically separate safety measure/adverse event reporting. Given the different patient numerator and denominator criteria we report each distinct adverse event (AE) measure separately within this record.
  Clinical decision support: Clinical decision support nudges within the electronic health record.
  The populations of patients monitored for adverse events varies depending on the numerator/denominator criteria for each separate safety measure/AE reported. Thus, the number of patients at risk varies by measure.
Arm/Group | Clinical Decision Support Intervention
All-Cause Mortality (participants affected / at risk) | 0/664
Serious Adverse Events (participants affected / at risk) | 0/664
Other Adverse Events (participants affected / at risk) | 0/664

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2019-06-06): https://cdn.clinicaltrials.gov/large-docs/89/NCT03704389/Prot_000.pdf